CLINICAL TRIAL: NCT04739969
Title: Rapid Acting Transcranial Magnetic Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor, Department of Psychiatry and Behavioral Sciences, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58807
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Depression
Keywords: transcranial magnetic stimulation; theta burst
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TBS-DLPFC (Active Comparator): The active group will receive theta-burst TMS stimulation.
  Interventions: Device: Active TBS-DLPFC
- Sham TBS-DLPFC (Sham Comparator): The sham group will receive sham theta-burst TMS stimulation.
  Interventions: Device: Sham TBS-DLPFC

INTERVENTIONS:
Device: Active TBS-DLPFC — Participants in the active stimulation group will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Soterix Neural Navigator neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro TMS system (MagVenture, Denmark).
  Arms: Active TBS-DLPFC
Device: Sham TBS-DLPFC — The parameters in the sham arm will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham TBS-DLPFC

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for treatment-resistant depression. In a double-blind, randomized, sham-controlled fashion, half the participants will receive accelerated theta-burst stimulation while half will receive sham treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been effective in real world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session, 5 days per week, for 4-8 weeks). Recently, we have pursued modifying the treatment parameters to reduce treatment times with an accelerated treatment paradigm with great preliminary success. This study aims to further study our accelerated protocol and examine changes in neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, between the ages of 22 and 65 at the time of screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening.

   Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
3. Currently diagnosed with Major Depressive Disorder (MDD) and meets criteria for a Major Depressive Episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
4. Medical records confirming a history of moderate to severe treatment-resistance as defined by a score of 7-14 on the Maudsley Staging Method (MSM 3).
5. MADRS score of ≥20 at screening (Visit 1).
6. TMS naive.
7. Access to ongoing psychiatric care before and after completion of the study.
8. Access to clinical rTMS after study completion.
9. Must be on a stable antidepressant therapeutic regimen for 6 weeks prior to study enrollment and agree to continue this regimen throughout the study period.
10. In good general health, as evidenced by medical history.
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
12. Agreement to adhere to Lifestyle Considerations throughout study duration.

Lifestyle Considerations:

* Abstain from becoming pregnant from the screening visit (Visit 1) until after the final study visit (Visit 13).
* Continue usual intake patterns of caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) without significant change for the duration of the study.
* Abstain from alcohol for at least 24 hours before the start of each MRI and TMS session.
* Participants who use tobacco products will be informed that use will be allowed only in between intervention sessions.

Exclusion Criteria:

1. Pregnancy
2. Primary psychiatric condition other than MDD requiring treatment except stable comorbid anxiety disorder
3. History of or current psychotic disorder or bipolar disorder
4. Severe borderline personality disorder.
5. Diagnosis of Intellectual Disability or Autism Spectrum Disorder
6. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
7. Urine screening test positive for illicit substances
8. Active suicidal ideation (defined as an MSSI > 8) or a suicide attempt (as defined by the C-SSRS) within the past one year
9. Any history of ECT (greater than 8 sessions) without meeting responder criteria
10. Recent (within 4 weeks of any clinical effect) or concurrent use of rapid acting antidepressant agent (i.e., ketamine or a course of ECT)
11. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
12. Untreated or insufficiently treated endocrine disorder.
13. Contraindication to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
14. Contraindication to MRI (ferromagnetic metal in their body)
15. Treatment with an investigational drug or other intervention within the study period
16. Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO)
17. Unstable symptoms between screening and baseline as defined by a ≥ 30% change in MADRS score.
18. Any other condition deemed by the PD to interfere with the study or increase risk to the participant

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rates of remission one month after treatment in the Montgomery-Åsberg Depression Rating Scale (MADRS) score. | Baseline, 1-month.
  The Montgomery-Åsberg Depression Rating Scale (MADRS), is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Remission is defined as MADRS ≤10.

SECONDARY OUTCOMES:
Rates of response one month after treatment in the Montgomery-Åsberg Depression Rating Scale (MADRS) score. | Baseline, 1-month.
  The Montgomery-Åsberg Depression Rating Scale (MADRS), is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Response is defined as a reduction of >/=50% of MADRS baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396